CLINICAL TRIAL: NCT02491164
Title: Exploratory Clinical Study of Intrapulmonary Microdosing of Gram-negative Optical Molecular Imaging BACterial Detection Probe
Brief Title: Exploratory Study of Intrapulmonary Microdosing of Gram-negative Optical Imaging Detection Probe
Acronym: BAC TWO
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BAC TWO
Record Dates: First submitted 2015-07-01; First posted 2015-07-07 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Respiratory Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BAC TWO administration (Experimental): All participants in this clinical study will be dosed on one occasion with BAC TWO. The final dosage will be 80 µg (± 25%).
  Interventions: Other: BAC TWO; Device: FE and Cellvizio viewer software

INTERVENTIONS:
Other: BAC TWO — BAC TWO administration
Device: FE and Cellvizio viewer software — Fibre based endomicroscopy to visualise fluorescent signal emitted by optical agents.

SUMMARY:
Critically ill patients are often ventilated in dedicated critical care units to provide respiratory support. Despite best practice patients can often develop a condition called adult respiratory distress syndrome (ARDS), which is characterised by deterioration in their respiratory function, and changes on chest x-ray. The correct management for ARDS is identifying the underlying condition causing the deterioration and identifying appropriate targeted therapy. One such cause is pneumonia, caused by a bacterial infection in the lungs of a ventilated patient. The patients may have been ventilated due to pneumonia but they may also develop pneumonia whilst ventilated. Ventilator associated pneumonia (VAP) has significant mortality.

Despite all the clinical and laboratory data at the investigators' disposal there remains great difficulty in the accurate diagnosis of pneumonia and therefore treatment is often given empirically. Therefore, there is an urgent clinical need for accurate methods to diagnose the presence of bacteria deep in the lung in ventilated critically ill patients. As such, the investigating team have developed and synthesised an imaging agent called BAC TWO. BAC TWO will be instilled directly into the lungs of 12 patients to assess whether it can label gram-negative bacteria in the human lung.

DETAILED DESCRIPTION:
The primary objective of this study is to deliver a BAC TWO microdose to 3 ventilated controls and 9 patients to assess the imaging parameters of BAC TWO over human autofluorescence and to assess if gram-negative bacteria can be detected in vivo in situ within the distal lung. The primary endpoint is to visualise the delivery of a microdose of BAC TWO and assess imaging parameters in;

* 3 mechanically ventilated patients to provide a control population (cohort 1)
* 6 bronchiectasis patients with predominant colonisation with gram-negative bacteria (cohort 2)
* 6 bronchiectasis patients with predominant colonisation with gram-positive bacteria (cohort 3)
* 3 patients with suspected pneumonia and pulmonary infiltrates in ICU (cohort 4)

For all cohorts, eligibility will be verified by a clinical trial physician after written informed consent has been obtained. For all cohorts, a bronchoscopy with lavage will be performed to harvest broncho-alveolar lavage fluid (BALF). Fibre-based endomicroscopy (FE) will be performed on up to three areas and up to 80μg (± 25%) in total of BAC TWO will be instilled in up to 3 sites.

Participants will be asked to provide additional blood and urine samples with the intention of examining for systemic uptake of the BAC TWO probe. Routine blood investigations will be performed 4-6 hours following the administration of BAC TWO. The completion of all assessments at 4-6 hours post dose marks the end of the participant's participation in this study unless there are ongoing adverse events requiring resolution. The primary aim will be measured during bronchoscopy and all routine investigations will have been completed 6 hours post dose.

ELIGIBILITY:
Inclusion Criteria:

All cohorts

* ≥ 16 years
* Attending consultant permission for bronchoscopy

Cohort 1

* Patients scheduled to undergo surgery under general anaesthesia
* Absence of acute or significant chronic lung disease as determined by the clinical suspicion of the attending medical team or of a medically qualified member of the study investigation team.
* Presence or scheduled presence of endo-tracheal tube.
* Capacity to provide informed consent

Cohort 2 and 3

* Patients with bronchiectasis with known microbiological predominance of gram-negative or gram-positive bacteria.
* Capacity to provide informed consent

Cohort 4

* Patients in the ICU with pulmonary infiltrates on radiological assessment
* Presence of invasive tracheal ventilation tube
* Provision of informed consent from the patient or their personal legal representative prior to any study related procedures.

Exclusion Criteria:

All cohorts

* Refusal for participation by attending consultant
* Any history of anaphylaxis or allergy to polymyxin-based antibiotics e.g. colomycin
* Significant coagulopathy, which causes bronchoscopy to be unsuitable, as determined by clinical co-investigator or the participant's attending consultant, using information which is routinely available
* Myocardial infarction in the preceding four weeks
* Women who are pregnant or are breastfeeding
* Receiving drugs that cause increased autofluorescence in the lung, specifically amiodorane and methotrexate

Cohort 4 only

* Inspired Oxygen Concentration (FiO2) >70%
* Positive End Expiratory Pressure (PEEP) >10cm
* Endotracheal tube (ETT) or tracheostomy internal diameter < 7mm
* Presence of pneumothorax
* Active bronchospasm
* Mean arterial pressure <65mmHg (millimeter of mercury) AND on vasopressor
* Platelet count < 50 x 109/L

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Imaging parameters of BAC TWO in the distal lung | up to 1 week post dose
  The main primary outcome measure is to visualise the delivery of BAC TWO in the distal lung of both ventilated controls and patients with gram-negative bronchiectasis, gram-positive bronchiectasis and pulmonary infiltrates through the measurement of fluorescence using FE and Cellvizio viewer software.

CONTACTS AND LOCATIONS:
Overall Officials: Kev Dhaliwal, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No